CLINICAL TRIAL: NCT07248813
Title: Effectiveness of an Additional Telerehabilitation Program Combined With Conventional Care on Functional Improvement in Patients With Chronic Low Back Pain at the Primary Care Level in the Mexican Institute of Social Security (IMSS): A Pragmatic Randomized Controlled Trial
Brief Title: Telerehabilitation Program to Improve Function in People With Chronic Low Back Pain Compared With Conventional Care
Acronym: TELEREHAB-LC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2025-1401-018
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Low Back Pain (Non-specific, Uncomplicated)
Keywords: TELEMEDICINE; Physical Therapy; Primary Care; Oswestry Disability Index; Rehabilitation Program; Telerehabilitation; Pragmatic Clinical Trial; Pain Management; Adherence
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to one of two parallel groups. The intervention group receives conventional care plus a six-week telerehabilitation program, while the control group receives conventional care only. Both groups are followed in parallel without crossover.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts are blinded to group allocation. Participants and care providers are not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation plus Conventional Care (Experimental): Participants in this group receive a six-week telerehabilitation program in addition to conventional medical care for chronic low back pain. The telerehabilitation program is delivered through the Moodle platform and includes educational videos, stretching and strengthening exercises based on Williams and McKenzie methods, core stabilization routines, relaxation techniques, and weekly virtual sessions. Conventional care includes physician consultations, analgesic treatment as needed, and ergonomic advice.
  Interventions: Behavioral: Telerehabilitation Program; Other: Conventional care
- Conventional Care Only (Active Comparator): Participants in this group receive standard medical care for chronic low back pain provided at IMSS primary care clinics. This includes physician consultations, pharmacologic management (analgesics, NSAIDs), ergonomic recommendations, and the institutional educational brochure on back hygiene and exercises. No telerehabilitation components are provided.
  Interventions: Other: Conventional care

INTERVENTIONS:
Behavioral: Telerehabilitation Program — A six-week telerehabilitation program provided in addition to conventional medical care for patients with chronic low back pain. The program is delivered through the Moodle platform and supported by WhatsApp communication. It includes five progressive modules with educational videos, stretching and strengthening exercises based on Williams and McKenzie methods, core stabilization and flexibility routines, and relaxation techniques adapted from Jacobson's progressive relaxation. Participants complete home-based exercises and one weekly virtual session, record their activities in logs, and receive feedback from the rehabilitation team.
  Arms: Telerehabilitation plus Conventional Care
Other: Conventional care — Standard medical care provided at IMSS primary care clinics for patients with chronic low back pain. It includes physician consultations, pharmacologic management as needed (analgesics, NSAIDs), ergonomic and posture advice, and the institutional educational brochure on back hygiene and exercises. No telerehabilitation components are included

SUMMARY:
The goal of this clinical trial is to evaluate whether an additional telerehabilitation program, combined with conventional care, can improve functional recovery in adults with chronic low back pain treated in primary care clinics of the Mexican Institute of Social Security (IMSS).

The main questions it aims to answer are:

* Does the telerehabilitation program lead to greater functional improvement, measured by the Oswestry Disability Index (ODI), compared with conventional care alone?
* Does the program reduce pain intensity and improve adherence and satisfaction among participants?

Researchers will compare patients receiving conventional care plus telerehabilitation with those receiving conventional care only to determine whether the digital intervention provides additional clinical benefits.

Participants will:

* Continue their usual medical care for chronic low back pain at IMSS clinics.
* Follow a 6-week telerehabilitation program delivered through an online platform, including educational videos, stretching and strengthening exercises, and weekly virtual check-ins.
* Complete baseline and post-intervention assessments of pain, disability, and satisfaction.

DETAILED DESCRIPTION:
Low back pain is the leading cause of musculoskeletal disability worldwide and represents one of the main reasons for medical consultation and work incapacity within the Mexican Institute of Social Security (IMSS). In Mexico, approximately 30 % of adults experience low back pain, and this condition is among the top ten causes of temporary work disability in the IMSS. Delays in referral to rehabilitation services often extend recovery time, increase institutional costs, and limit patients' functional reintegration.

Telerehabilitation has emerged as a promising alternative to improve accessibility, continuity of care, and adherence in musculoskeletal conditions. It allows the delivery of structured therapeutic exercise programs and education modules through digital platforms, reducing logistical barriers and waiting times. However, evidence on its clinical effectiveness in public healthcare systems, particularly in pragmatic real-world settings such as IMSS primary care units, remains scarce.

This pragmatic randomized controlled clinical trial aims to evaluate the effectiveness and feasibility of an additional telerehabilitation program combined with conventional care, compared with conventional care alone, in improving functional outcomes in adults with chronic non-specific low back pain. The study is conducted at Family Medicine Unit No. 69 (UMF 69) in Texcoco, State of Mexico, which provides first-level care for musculoskeletal disorders.

Participants aged 18-60 years with clinically diagnosed chronic low back pain (duration ≥ 12 weeks) are recruited consecutively from IMSS outpatient consultations. After obtaining informed consent, eligible participants are randomly assigned in a 1:1 ratio to either the intervention group (telerehabilitation + conventional care) or the control group (conventional care only), using a computer-generated randomization list with concealed allocation. Outcome assessors and data analysts remain blinded to group assignment.

The telerehabilitation program consists of a six-week structured protocol delivered through the Moodle platform and supported by WhatsApp communication. It includes five progressive modules that integrate:

Education on disease understanding and self-management.

Spine hygiene and ergonomic recommendations.

Physical therapy exercises based on Williams and McKenzie methods.

Core strengthening and stretching routines.

Relaxation and breathing techniques adapted from Jacobson's progressive relaxation.

Weekly asynchronous educational videos are complemented by one live (synchronous) virtual session per week, promoting interaction and motivation. Participants record their daily exercises and pain levels in printed or digital logs, which are reviewed weekly. Adherence is monitored by login frequency, participation in virtual sessions, and completion of exercise diaries.

The control group receives conventional medical management from family physicians, which may include pharmacologic therapy (analgesics, NSAIDs), ergonomic advice, and distribution of the institutional educational brochure on back hygiene and exercise (Williams series). This reflects the routine standard of care in IMSS primary care settings and intentionally preserves clinical variability to enhance external validity.

The primary outcome is functional improvement measured by the Oswestry Disability Index (ODI), comparing baseline and six-week scores between groups. The secondary outcomes include pain intensity (Visual Analogue Scale, VAS), time to functional recovery, adherence to the intervention, and participant satisfaction. The study hypothesizes that the telerehabilitation program will achieve a ≥ 10-point greater reduction in ODI scores (the minimal clinically important difference) compared with conventional care.

A total of 200 participants (100 per group) will be included, accounting for an expected 40 % attrition rate and ensuring sufficient power (80 %) to detect the predefined difference. Data will be analyzed under the intention-to-treat principle using ANCOVA adjusted for confounders (age, body-mass index, comorbidities, and physical activity level). Complementary logistic regression will assess the proportion of participants achieving clinically meaningful improvement.

This pragmatic design reflects real-world clinical practice and aims to generate evidence directly applicable to IMSS settings. The study's feasibility is supported by existing infrastructure, including access to the IMSS Moodle platform, telecommunication tools, and trained personnel in rehabilitation medicine.

The trial is classified as greater-than-minimal risk under Mexican health regulations because it involves an experimental therapeutic modality; however, it is considered low physical risk since all exercises correspond to standard rehabilitation practice. Ethical approval was granted by the Local Research and Ethics Committee No. 1401 (IMSS), and all participants provide written informed consent. Participant confidentiality is protected according to Mexican data protection law and institutional guidelines.

The study adheres to the Declaration of Helsinki, the Belmont Report, and the General Health Law on Research for Human Subjects (Mexico). The trial's oversight and safety monitoring are performed by the principal investigator and the local ethics board; no independent Data Monitoring Committee is established, given the minimal risk of the intervention.

If proven effective, this program could provide an accessible, low-cost, and scalable rehabilitation strategy within primary care, reducing disability, improving patient satisfaction, and optimizing healthcare resources. The findings will support institutional decision-making for the gradual implementation of telerehabilitation across IMSS facilities and contribute to national strategies for strengthening rehabilitation services, as recommended by the World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 60 years of age.
* Clinical diagnosis of chronic non-specific low back pain (duration ≥ 12 weeks).
* Pain intensity ≥ 3 on the Visual Analogue Scale (VAS) at baseline.
* Enrolled as beneficiaries of the Mexican Institute of Social Security (IMSS) and receiving care at a primary care clinic.
* Access to a smartphone or computer with internet connection.
* Ability to read and understand written instructions in Spanish.
* Willingness to participate and provide written informed consent.

Exclusion Criteria:

* Specific causes of low back pain (e.g., fractures, tumors, infections, inflammatory or rheumatic diseases).
* Neurological deficits suggestive of radiculopathy or myelopathy.
* Pregnancy.
* Severe psychiatric or cognitive disorders that limit participation.
* Recent spinal surgery (within the last 6 months).
* Participation in another rehabilitation or exercise program for low back pain within the previous 3 months.
* Any medical condition that contraindicates physical exercise, as determined by the treating physician.

The upper age limit of 60 years was established to minimize confounding factors related to advanced degenerative joint disease. Individuals older than 60 frequently present radiographic or clinical signs of grade III or higher lumbar osteoarthritis, which may produce chronic pain and functional limitation independent of the intervention. Including these participants could obscure the true effect of the telerehabilitation program on functional improvement and pain reduction in patients with non-specific chronic low back pain.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Functional improvement measured by the Oswestry Disability Index (ODI) | Baseline and 6 weeks after randomization
  Change in functional disability score assessed using the validated Spanish version of the Oswestry Disability Index (ODI). The scale measures the degree of disability related to low back pain across 10 domains (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment). Scores range from 0 (no disability) to 100 (maximum disability).

SECONDARY OUTCOMES:
Pain Intensity | Baseline and 6 weeks after randomization
  Change in pain intensity measured using the Visual Analogue Scale (VAS). Participants rate their average pain over the previous week on a 10 cm line ranging from 0 (no pain) to 10 (worst imaginable pain).
Participant Satisfaction | At the end of the 6-week intervention
  Satisfaction with the intervention measured using a Likert-type questionnaire (1-5 scale) evaluating accessibility, clarity of information, usefulness of exercises, and overall satisfaction with care.
Time to Functional Recovery | Up to 6 weeks after baseline
  Time (in days) from enrollment to the first report of ≥10-point reduction in ODI score, representing the minimal clinically important difference (MCID).

OTHER OUTCOMES:
Adherence to the Telerehabilitation Program | Throughout the 6-week intervention period
  Percentage of participants who complete at least 80% of the telerehabilitation sessions and daily exercise logs. Adherence is tracked through Moodle platform activity, attendance at virtual sessions, and completion of exercise diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Arlette R. Ordoñez Flores, MD, MSc, Principal Investigator — Instituto Mexicano del Seguro Social; David R. Mejía, MD, PhD, Study Chair — Instituto Mexicano del Seguro Social; José de Jesús R. Sánchez, MD, PhD, Study Chair — Hospital General de México Eduardo Liceaga; Rodolfo P. Almazán, PhD, Study Chair — National Polytechnic Institute, Mexico
Locations (1):
- Family Medicine Unit No. 69, Mexican Institute of Social Security (IMSS), México, Texcoco, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains confidential health information owned by the Mexican Institute of Social Security (IMSS). Data sharing is restricted by institutional and national regulations on personal data protection. Only aggregated and anonymized results will be available upon reasonable request and after institutional approval.

REFERENCES:
- [Background] Simsek A, Ulger O. Effectiveness of telerehabilitation exercises in low back pain: a systematic review. Ir J Med Sci. 2025 Oct;194(5):1903-1913. doi: 10.1007/s11845-025-04051-x. Epub 2025 Aug 13. PMID 40802146
- [Background] Villatoro-Luque FJ, Rodriguez-Almagro D, Aibar-Almazan A, Fernandez-Carnero S, Pecos-Martin D, Ibanez-Vera AJ, Castro-Martin E, Achalandabaso-Ochoa A. Telerehabilitation for the treatment in chronic low back pain: A randomized controlled trial. J Telemed Telecare. 2025 Jun;31(5):637-646. doi: 10.1177/1357633X231195091. Epub 2023 Aug 30. PMID 37649362
- [Background] Lara-Palomo IC, Gil-Martinez E, Ramirez-Garcia JD, Capel-Alcaraz AM, Garcia-Lopez H, Castro-Sanchez AM, Antequera-Soler E. Efficacy of e-Health Interventions in Patients with Chronic Low-Back Pain: A Systematic Review with Meta-Analysis. Telemed J E Health. 2022 Dec;28(12):1734-1752. doi: 10.1089/tmj.2021.0599. Epub 2022 May 9. PMID 35532971
- [Background] Sivertsson J, Sernert N, Ahlund K. Exercise-based telerehabilitation in chronic low back pain - a scoping review. BMC Musculoskelet Disord. 2024 Nov 23;25(1):948. doi: 10.1186/s12891-024-07952-7. PMID 39580408
- See also: World Health Organization - Digital Health and Telemedicine. Offers information on digital health strategies, including telemedicine and remote rehabilitation, endorsed by the World Health Organization. — https://www.who.int/health-topics/digital-health#tab=tab_1